CLINICAL TRIAL: NCT06875687
Title: Effects of a Prostaglandin Analog-Based Eyelash Serum on Ocular Surface Integrity and Tear Film Stability: A Prospective Interventional Study
Brief Title: Prostaglandin Analog Eyelash Serum and Ocular Surface Health: A Prospective Study
Acronym: EYESERUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, José-María Sánchez-González, Head of Vision Science Research Group, University of Seville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: USeville_2025_02
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
Keywords: Prostaglandin analog; Eyelash growth; Ocular surface; Tear film stability; Ophthalmic safety
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional study evaluating the effects of a prostaglandin analog-based eyelash serum on ocular surface integrity, tear film stability, and eyelash growth over six weeks. All participants applied the serum daily, and clinical assessments were performed at baseline and post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostaglandin Analog-Based Eyelash Serum Group (Experimental): This study arm consists of healthy female participants who applied a prostaglandin analog-based eyelash serum once daily to the upper eyelid margin for six weeks. The study evaluated changes in ocular surface integrity, tear film stability, and eyelash growth. Clinical assessments were performed at baseline and post-treatment, including measurements of tear film parameters, ocular hyperemia, and intraocular pressure.
  Interventions: Other: Prostaglandin Analog-Based Eyelash Serum

INTERVENTIONS:
Other: Prostaglandin Analog-Based Eyelash Serum — This intervention consists of a prostaglandin analog-based eyelash serum applied once daily to the upper eyelid margin for six weeks. The serum contains dechloro dihydroxy difluoro ethylcloprostenolamide (DDDE), a prostaglandin analog known to promote eyelash growth. The formulation also includes panax ginseng root extract, urtica dioica extract, panthenol, niacinamide, and biotinoyl tripeptide-1, which contribute to hair follicle nourishment. The study evaluates its effects on ocular surface integrity, tear film stability, and eyelash growth.
  Other Names: Eyelash Growth Serum; Prostaglandin Analog Eyelash Enhancer

SUMMARY:
This prospective interventional study investigates the effects of a prostaglandin analog-based eyelash serum on ocular surface integrity, tear film stability, and eyelash growth over six weeks. Nineteen healthy female participants applied the serum daily, with clinical assessments performed at baseline and post-treatment. The study adhered to ethical guidelines, and parameters such as tear film stability, tear volume, ocular hyperemia, and eyelash characteristics were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals aged 18 to 30 years.
* Corrected distance visual acuity (CDVA) of 0.10 LogMAR or better in both eyes.
* Fitzpatrick skin type III or lower.
* No active dermatological conditions affecting the periocular area.
* Regular use of cosmetic products (e.g., mascara, eyeliner, or eyeshadow) with no history of intolerance.
* Willingness and ability to follow the serum application protocol for six weeks.

Exclusion Criteria:

* History or diagnosis of dry eye disease or other ocular surface disorders.
* Previous ocular surgery, trauma, or systemic conditions affecting ocular surface function.
* Use of topical or systemic medications that could impact tear film stability.
* Documented hypersensitivity or allergic reactions to cosmetic or ophthalmic products.
* Presence of eyelid disorders that could interfere with eyelash growth (e.g., blepharitis, trichiasis).
* Use of growth-enhancing serums within the past three months.
* Pregnancy or breastfeeding at the time of enrollment.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Tear Film Stability (A-NIBUT) After Six Weeks of Eyelash Serum Application | Baseline and after six weeks of serum application
  Assessment of average non-invasive tear break-up time (A-NIBUT) as an indicator of tear film stability before and after six weeks of daily prostaglandin analog-based eyelash serum application. A-NIBUT is measured using the Firefly S390I slit lamp (MediWorks, Suzhou, China), with lower values indicating increased tear film instability.

SECONDARY OUTCOMES:
Change in Tear Volume (Tear Meniscus Height - TMH) After Six Weeks | Baseline and after six weeks
  Measurement of tear meniscus height (TMH) before and after six weeks of eyelash serum application using the Firefly S390I slit lamp to assess changes in aqueous tear volume. Lower TMH values indicate a reduction in tear production.
Change in Ocular Hyperemia (Conjunctival and Ciliary Hyperemia) After Six Weeks | Baseline and after six weeks
  Evaluation of temporal conjunctival hyperemia (TCOH) and temporal ciliary hyperemia (TCIH) using digital image analysis. An increase in hyperemia suggests a vasodilatory response to the serum.
Change in Eyelash Length and Thickness After Six Weeks | Baseline and after six weeks
  Measurement of eyelash length and thickness before and after six weeks using caliper software on the Firefly S390I slit lamp to determine the efficacy of the serum in promoting eyelash growth.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and ethical considerations. The collected data include sensitive ocular health parameters, and sharing such data could compromise participant confidentiality. However, aggregated data and study results will be available upon reasonable request for academic and research purposes.

REFERENCES:
- [Background] Alonso MR, Damonte SP, Anesini C. Jarilla-Coffea extract: a natural cosmetic product that improves eyelash and eyebrow growth in women. Clin Cosmet Investig Dermatol. 2019 Jan 9;12:47-55. doi: 10.2147/CCID.S182497. eCollection 2019. PMID 30666142
- [Background] Fernandez-Gonzalez P, Truchuelo-Diez MT, Gomez-Sanchez MJ. Open clinical trial evaluating the efficacy of a novel eyelash growth enhancer with peptides and glycosaminoglycans. J Cosmet Dermatol. 2024 Jun;23(6):2170-2180. doi: 10.1111/jocd.16265. Epub 2024 Apr 4. PMID 38572527
- [Background] Sachdev M, Velugotla K, Revanker S, Somasekhar G. An Open-label, Single-center, Safety and Efficacy Study of Eyelash Polygrowth Factor Serum. J Clin Aesthet Dermatol. 2020 Feb;13(2):61-66. Epub 2020 Feb 1. PMID 32308787
- [Background] Kim YK, Woo IS, Park CG, Kim A, Choi JD, Son KH, Han KM. Green extraction of prostaglandin analogs in cosmetics using deep eutectic solvents and detection via LC-MS/MS. J Chromatogr A. 2025 Jan 4;1739:465516. doi: 10.1016/j.chroma.2024.465516. Epub 2024 Nov 13. PMID 39579545
- [Background] Baiyasi M, St Claire K, Hengy M, Tur K, Fahs F, Potts G. Eyelash serums: A comprehensive review. J Cosmet Dermatol. 2024 Jul;23(7):2328-2344. doi: 10.1111/jocd.16278. Epub 2024 Mar 12. PMID 38475901